CLINICAL TRIAL: NCT05587998
Title: A Randomized, Double-blind, Placebo-controlled, Fixed Sequence Study to Assess the Effect on Respiratory Drive of Multiple Doses of AZD4041 When Co-administered With a Single Dose of Morphine in Healthy Recreational Opioid Users
Brief Title: A Study to Assess the Effect of AZD4041 on Respiratory Drive in Recreational Opioid Users.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D7460C00003
Record Dates: First submitted 2022-09-21; First posted 2022-10-20 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Morphine then AZD4041 then Morphine + AZD4041 (Experimental): Participants will receive a single intravenous (IV) dose of morphine Dose Level 1 on Day 1. From Day 2 to Day 15, participants will receive an oral dose of AZD4041 Dose Level 1, once daily for 14 consecutive days. On Day 15, participants will receive an oral dose of AZD4041 Dose Level 1 in combination with a single IV dose of morphine Dose Level 1.
  Interventions: Drug: Morphine; Drug: AZD4041
- Morphine then Placebo then Morphine + Placebo (Placebo Comparator): Participants will receive a single IV dose of morphine Dose Level 1 on Day 1. From Day 2 to Day 15, participants will receive an oral dose of placebo matched to AZD4041, once daily for 14 consecutive days. On Day 15, participants will receive an oral dose of placebo matched to AZD4041 in combination with a single IV dose of morphine Dose Level 1.
  Interventions: Drug: Morphine; Other: Placebo

INTERVENTIONS:
Drug: Morphine — Participants will receive IV dose of Morphine as stated in arm description.
  Other Names: Duramorph PF®
Drug: AZD4041 — Participants will receive oral doses of AZD4041 as stated in arm description.
  Other Names: No other names
  Arms: Morphine then AZD4041 then Morphine + AZD4041
Other: Placebo — Participants will receive oral doses of placebo as stated in arm description.
  Other Names: No other names
  Arms: Morphine then Placebo then Morphine + Placebo

SUMMARY:
This is a Phase 1, single-centre, randomized, double-blind, placebo-controlled, 2 fixed sequences, multiple dose study in healthy male and/or female recreational opioid users.

This study is being primarily conducted to assess the effect on respiratory drive of morphine administered after multiple doses of AZD4041 compared to morphine administered alone in healthy recreational opioid users.

The study will include up to 44 participants who will be randomized to either AZD4041 and morphine (28 participants) or placebo and morphine (16 participants). This is to ensure completion of at least 36 participants (24 AZD4041 + morphine, and 12 Placebo + morphine on Day 15).

The total study duration will be up to 54 days (including screening) per participant.

ELIGIBILITY:
Inclusion Criteria:

1. Recreational opioid user, not currently considered to have moderate or severe substance use disorder for opioids (based on the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition [DSM-5] criteria) and has experience with opioid use for non-therapeutic purposes (ie, for psychoactive effects) on at least 10 occasions in their lifetime and at least 1 occasion in the last 12 weeks prior to screening.
2. Provision of signed and dated informed consent form (ICF) prior to the initiation of any protocol-specific procedures.
3. Stated willingness to comply with all study procedures and availability for the duration of the study.
4. Healthy adult male or female, 18 to 55 years of age, inclusive, prior to the first study drug administration.
5. Body mass index (BMI) within 18.0 kg/m^2 to 35.0 kg/m^2, inclusive, and body weight at least 50 kg at screening.
6. A female study participant of non-childbearing potential must meet 1 of the following criteria:

(1) Physiological postmenopausal status, defined as the following:

1. absence of menses for at least 1 year prior to the first study drug administration (without an alternative medical condition); and
2. Follicle stimulating hormone (FSH) levels ≥ 40 mIU/mL at screening

   AND/OR

   (2) Surgical sterile, defined as those who have had hysterectomy, bilateral oophorectomy and/or bilateral salpingectomy, or bilateral tubal ligation. Women who are surgically sterile must provide documentation of the procedure by an operative report, ultrasound, or other verifiable documentation.

   7. If male, must agree to use a highly effective method of contraception when engaging in sexual activity and must not donate sperm during the study and for at least 4 months (120 days) after the last dose of study medication.

   8. Healthy in the opinion of an Investigator, as determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs, SpO2, respiratory rate, or clinical laboratory (including hematology, coagulation, clinical chemistry, urinalysis, and serology [screening visit only]) at screening visit and/or prior to the first study drug administration.

   Exclusion Criteria:
   1. Female who is pregnant according to the pregnancy test at screening or prior to the first study drug administration.
   2. Male participants with a history of oligospermia or azoospermia or any other disorder of the reproductive system.
   3. Male participants who are undergoing treatment or investigation for infertility.
   4. History of moderate or severe substance or alcohol use disorder (excluding nicotine and caffeine) within the past 2 years, as defined by the DSM-5.
   5. History of any significant psychiatric disorder according to the criteria of the DSM-5 which, in the opinion of the Investigator, could be detrimental to participant safety or could compromise study data interpretation.
   6. History of significant hypersensitivity to AZD4041, morphine and/or other opioids, naloxone, or any related products (including excipients of the study formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
   7. History of any significant disease, including [but not necessarily limited to] significant hepatic, renal, cardiovascular, pulmonary, hematologic, neurological, psychiatric, gastrointestinal, endocrine, immunologic, ophthalmologic, or dermatologic disease of any etiology (including infections) identified at screening.
   8. Presence or history of significant gastrointestinal, liver or kidney disease, or any other condition [including those that may result from surgery] that is known to interfere with drug absorption, distribution, metabolism, or excretion, or known to potentiate or predispose to undesired effects.
   9. SpO2 below 95% at screening or prior to first study drug administration.
   10. Any abnormal vital signs, after no less than 5 minutes rest (supine position), as defined in the list below, at screening and/or prior to the first study drug administration. Out of range test may be repeated once for each visit at the discretion of the Investigator.

       1. Systolic Blood Pressure (BP) < 90 mmHg or > 140 mmHg
       2. Diastolic BP < 50 mmHg or > 90 mmHg
       3. Heart Rate (HR) < 45 or > 90 beats per minute (bpm)
   11. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG, which in the Investigator's opinion, may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol-defined primary lead, or left ventricular hypertrophy at screening or prior to the first study drug administration (out of range test may be repeated once for each visit at the discretion of the Investigator).
   12. Prolonged QT interval corrected for HR using Fridericia's formula (QTcF) > 450 ms at screening or prior to first study drug administration.
   13. Shortened QTcF < 340 ms at screening or prior to first study drug administration.
   14. Family history of long QT syndrome.
   15. ECG interval measured from the onset of the P wave to the onset of the QRS complex (PR [PQ]) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular preexcitation) at screening or prior to first study drug administration.
   16. PR (PQ) interval prolongation (> 220 ms), persistent or intermittent second (Wenckebach block while asleep is not exclusive) or third degree atrioventricular (AV) block, or AV dissociation at screening or prior to first study drug administration.
   17. Persistent or intermittent complete bundle branch block, incomplete bundle branch block, or intraventricular conduction delay with ECG interval measured from the onset of the QRS complex to the J point (QRS) > 110 ms. Participants with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of ventricular hypertrophy or preexcitation at screening or prior to first study drug administration.
   18. In the predose 24-hour telemetry, presence of ≥ 10 ventricular premature contractions (VPCs) during 1 hour, or ≥ 100 VPCs during 24 hours of telemetry, or any occurrence of paired VPCs (ventricular couplets) or other repetitive ventricular rhythms, including non-sustained or sustained (> 30 second duration), slow (< 100 bpm), or fast (≥ 100 bpm) ventricular tachycardias.
   19. Any clinically significant illness in the 28 days prior to the first study drug administration.
   20. Heavy smoker (> 20 cigarettes per day) and/or is unable to abstain from smoking or unable to abstain from the use of prohibited nicotine containing products for at least 1 hour before and at least 6 hours after study drug administration (including e-cigarettes, pipes, cigars, chewing tobacco, nicotine topical patches, nicotine gum, or nicotine lozenges).
   21. Regularly consumes excessive amounts of caffeine or xanthines within 30 days prior to screening, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day.
   22. History of suicidal ideation within 1 year of screening (score of 4 or 5 as per the C-SSRS) or any suicidal behavior (as per C-SSRS) within 2 years of screening, or is currently at risk of suicide in the opinion of an Investigator.
   23. Positive test result for alcohol and/or drugs of abuse upon admission on Day -1. Participants with positive marijuana results at admission may be rescheduled at the discretion of an Investigator. If Tetrahydrocannabinol is positive at admission, a cannabis intoxication evaluation will be done by an Investigator and participants may be permitted to continue in the study at the discretion of an Investigator. Other positive test results should be reviewed to determine if the participant may be rescheduled, in the opinion of an Investigator.
   24. Positive test results for Human Immunodeficiency Virus (HIV)-1/HIV-2 Antibodies, Hepatitis B surface Antigen (HBsAg) or Hepatitis C Virus Antibody (HCVAb).
   25. Any other clinically significant abnormalities in laboratory test results at screening that would, in the opinion of an Investigator, increase the participant's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data.
   26. Treatment with an investigational drug within 30 days or 5 times the half-life (whichever is longer) prior to screening.
   27. Use of any prescription drugs (with the exception of hormone replacement therapy) in the 14 days prior to the first study drug administration, that in the opinion of an Investigator would put into question the status of the participant as healthy.
   28. Use of St. John's wort in the 28 days prior to the first study drug administration.
   29. Use of over-the-counter (OTC) products (including herbal preparations and supplements) within 7 days prior to the first study drug administration, with the exception of ibuprofen or acetaminophen.
   30. Donation of plasma in the 7 days prior to the first study drug administration.
   31. Donation of 1 unit of blood to American Red Cross or equivalent organization or donation of over 500 mL of blood in the 56 days prior to the first study drug administration.
   32. Is, in the opinion of an Investigator or designee, considered unsuitable or unlikely to comply with the Study Protocol for any reason.
   33. Poor venous access at screening, as judged by an Investigator.
   34. Use of any prescribed or nonprescribed oral and topical inhibitors/inducers of CYP3A4 (including shampoo).
   35. Is an AstraZeneca or study site employee or their close relatives.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, MD, Principal Investigator — Altasciences Company Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7460C00003&attachmentIdentifier=97f9d49c-a7f0-4b4a-bbbf-6096be8cd888&fileName=azd4041-d7460c00003-synopsis-redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Started | 29 | 16
Treated | 26 | 15
Completed | 25 | 13
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Not treated | 3 | 1
Not completed — Non-compliance with study procedures | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of morphine.
Groups:
- Morphine Then AZD4041 Then Morphine + AZD4041: Participants will receive a single IV dose of morphine Dose Level 1 on Day 1. From Day 2 to Day 15, participants will receive an oral dose of AZD4041 Dose Level 1, once daily for 14 consecutive days. On Day 15, participants will receive an oral dose of AZD4041 Dose Level 1 in combination with a single IV dose of morphine Dose Level 1.
- Total: Total of all reporting groups
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo | Total
Number analyzed (Participants) | 26 | 15 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.2 (6.76) | 34.8 (5.75) | 33.8 (6.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 23 | 14 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 23 | 15 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 12 | 31
  White | 7 | 3 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Increased End-tidal Carbon Dioxide (EtCO2) of at Least 10 mmHg Compared to Baseline or > 50 mmHg on Day 1
Description: ETCo2 measurement is performed in the clinical pharmacology setting studies for the evaluation of respiratory function. EtCO2 is monitored and measured using a standardized methodology and configuration using MICROSREAM^TM consumables to sample gas via nasal cannulae and the CAPNOSTREAM^TM20P bedside monitor according to Altasciences SOP on Capnography. Using this configuration, for the spontaneously breathing healthy volunteer participant, baseline EtCO2 measurements is expected to fall within the range of 34 to 48 mmHg. An increase in EtCO2 is defined as an increase of at least 10 mmHg compared to baseline or > 50 mmHg (sustained for at least 30 seconds). Number of participants with increased EtCO2 of at least 10 mmHg compared to baseline or > 50 mmHg on Day 1 are reported.
Time Frame: Day 1
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Increased End-tidal Carbon Dioxide (EtCO2) of at Least 10 mmHg Compared to Baseline or > 50 mmHg on Day 15
Description: ETCo2 measurement is performed in the clinical pharmacology setting studies for the evaluation of respiratory function. EtCO2 is monitored and measured using a standardized methodology and configuration using MICROSREAM^TM consumables to sample gas via nasal cannulae and the CAPNOSTREAM^TM20P bedside monitor according to Altasciences SOP on Capnography. Using this configuration, for the spontaneously breathing healthy volunteer participant, baseline EtCO2 measurements is expected to fall within the range of 34 to 48 mmHg. An increase in end tidal carbon dioxide (EtCO2) is defined as an increase of at least 10 mmHg compared to baseline or > 50 mmHg (sustained for at least 30 seconds). Number of participants with increased EtCO2 of at least 10 mmHg compared to baseline or > 50 mmHg on Day 15 are reported.
Time Frame: Day 15
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Participants | 2 | 1

3. Primary Outcome: Number of Participants With Reduction in Blood Oxygen Saturation (SpO2) to < 92% on Day 1
Description: A reduction in SpO2 is defined as a reduction from baseline to < 92% (sustained for at least 30 seconds). Number of participants with reduction in SpO2 to < 92% on Day 1 are reported.
Time Frame: Day 1
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Reduction in Blood Oxygen Saturation (SpO2) to < 92% on Day 15
Description: A reduction in SpO2 is defined as a reduction from baseline to < 92% (sustained for at least 30 seconds). Number of participants with reduction in SpO2 to < 92% on Day 15 are reported.
Time Frame: Day 15
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Participants | 1 | 0

5. Secondary Outcome: Time to Reduction in SpO2 to < 92%
Description: Mean time to reduction from baseline in SpO2 to < 92% (sustained for at least 30 seconds) is reported.
Time Frame: Day 1 and Day 15
Population: The safety population included all participants who received at least 1 dose of morphine. Number of participants analyzed (N) denotes only those participants who had reduction in SpO2 to < 92% (sustained for at least 30 seconds). On Day 1, number of participants with reduction in SpO2 to < 92% (sustained for at least 30 seconds) was 0.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 1 | 0
Hours
  Day 1: number analyzed (Participants) | 0 | 0
  Day 15 | 0.986 (NA) — Since, there was only one participant evaluable in this arm, standard deviation is not applicable. |

6. Secondary Outcome: Duration of Reduction in SpO2 to < 92%
Description: Mean duration of reduction from baseline in SpO2 to < 92% (sustained for at least 30 seconds) is reported.
Time Frame: Day 1 and Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 1 | 0
Minutes
  Day 1: number analyzed (Participants) | 0 | 0
  Day 15 | 1.083 (NA) — Since, there was only one participant evaluable in this arm, standard deviation is not applicable. |

7. Secondary Outcome: Post-dose Reduction of SpO2 Adjusted for Baseline
Description: Maximum post-dose reduction of SpO2 adjusted for baseline is reported.
Time Frame: Day 1, Day 8, and Day 15
Population: The safety population included all participants who received at least 1 dose of morphine. Here, number analyzed (n) denotes those participants who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Percent Reduction in SpO2
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Percent Reduction in SpO2
  Day 1 | 3.775 (1.5019) | 3.256 (1.6150)
  Day 8: number analyzed (Participants) | 25 | 14
  Day 8 | 3.286 (1.7564) | 2.751 (1.7650)
  Day 15: number analyzed (Participants) | 25 | 13
  Day 15 | 3.366 (2.3449) | 2.757 (1.7037)

8. Secondary Outcome: Post-dose SpO2
Description: Mean post-dose SpO2 is reported.
Time Frame: Day 15
Population: The safety population included all participants who received at least 1 dose of morphine. Number of participants analyzed (N) denotes the number of participants who were evaluable for the specified outcome measure.
Measure: Mean (Standard Deviation); unit: Percent SpO2
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 25 | 13
Percent SpO2 | 96.990 (1.6167) | 97.900 (1.2076)

9. Secondary Outcome: Time to Each Increased EtCO2 Episode of at Least 10 mmHg Compared to Baseline or > 50 mmHg
Description: Mean time to each increased EtCO2 episode of at least 10 mmHg compared to baseline or > 50 mmHg (sustained for at least 30 seconds) is reported.
Time Frame: Day 1 and Day 15
Population: The safety population included all participants who received at least 1 dose of morphine. Number of participants analyzed (N) denotes those participants who had EtCO2 of at least 10 mmHg compared to baseline or > 50 mmHg (sustained for at least 30 seconds). On Day 1, number of participants with increased EtCO2 of at least 10 mmHg compared to baseline or > 50 mmHg (sustained for at least 30 seconds) was 0.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 2 | 1
Hours
  Day 1: number analyzed (Participants) | 0 | 0
  Day 15 | 2.812 (1.6494) | 2.083 (NA) — Since, there was only one participant evaluable in this arm, standard deviation is not applicable.

10. Secondary Outcome: Duration of Each Increased EtCO2 Episode of at Least 10 mmHg Compared to Baseline or > 50 mmHg
Description: Mean duration of each increased EtCO2 episode of at least 10 mmHg compared to baseline or > 50 mmHg (sustained for at least 30 seconds) is reported.
Time Frame: Day 1 and Day 15
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 2 | 1
Minutes
  Day 1: number analyzed (Participants) | 0 | 0
  Day 15 | 8.202 (6.8859) | 0.750 (NA) — Since, there was only one participant evaluable in this arm, standard deviation is not applicable.

11. Secondary Outcome: Post-dose Increase in EtCO2 Adjusted for Baseline
Description: Maximum post-dose increase in EtCO2 adjusted for baseline is reported.
Time Frame: Day 1, Day 8, and Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
mmHg
  Day 1 | 6.501 (1.9432) | 7.177 (1.6955)
  Day 8: number analyzed (Participants) | 25 | 14
  Day 8 | 3.141 (2.8440) | 3.452 (2.1808)
  Day 15: number analyzed (Participants) | 25 | 13
  Day 15 | 7.261 (2.5220) | 7.462 (1.9624)

12. Secondary Outcome: Post-dose EtCO2
Description: Mean post-dose EtCO2 is reported.
Time Frame: Day 15
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 25 | 13
mmHg | 41.870 (2.8188) | 40.923 (2.4410)

13. Secondary Outcome: Number of Participants With Reduced Respiratory Rate (RR) of < 6 Breaths/Min
Description: Number of participants with RR of < 6 breaths/min (sustained for at least 30 seconds) are reported.
Time Frame: Day 1, Day 8, and Day 15
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Participants | 0 | 0

14. Secondary Outcome: Time to Each Reduced Respiratory Rate Episode of < 6 Breaths/Min
Description: Mean time to each reduced respiratory rate episode of < 6 breaths/min (sustained for at least 30 seconds) is reported.
Time Frame: Day 1, Day 8, and Day 15
Population: The safety population included all participants who received at least 1 dose of morphine. Number of participants with RR of < 6 breaths/min (sustained for at least 30 seconds) was 0.
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Duration of Each Reduced Respiratory Rate Episode of < 6 Breaths/Min
Description: Mean duration of each reduced respiratory rate episode of < 6 breaths/min (sustained for at least 30 seconds) is reported.
Time Frame: Day 1, Day 8, and Day 15
Population: as for outcome 14
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Post-dose Decrease in RR Adjusted for Baseline
Description: Maximum post-dose decrease in RR adjusted for baseline is reported.
Time Frame: Day 1, Day 8, and Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Breaths/min
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Breaths/min
  Day 1 | 4.852 (1.7684) | 5.523 (2.2649)
  Day 8: number analyzed (Participants) | 25 | 14
  Day 8 | 4.133 (2.5477) | 4.667 (2.1252)
  Day 15: number analyzed (Participants) | 25 | 13
  Day 15 | 5.133 (2.4346) | 6.116 (2.2576)

17. Secondary Outcome: Post-dose RR
Description: Mean post-dose RR is reported.
Time Frame: Day 15
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Breaths/minute
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 25 | 13
Breaths/minute | 13.577 (2.0284) | 13.477 (2.7037)

18. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through end of study (Day 24)
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Participants
  Any TEAEs | 26 | 14
  Any TESAEs | 0 | 0

19. Secondary Outcome: Number of TEAEs
Description: The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. Here, Number of TEAEs are reported.
Time Frame: Day 1 through end of study (Day 24)
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Number; unit: Events
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Events | 134 | 102

20. Secondary Outcome: Number of TEAEs by Severity
Description: The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. Here, number of TEAEs by severity (mild, moderate, or severe) are reported.
Time Frame: Day 1 through end of study (Day 24)
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Number; unit: Events
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Events
  Mild | 129 | 99
  Moderate | 5 | 3
  Severe | 0 | 0

21. Secondary Outcome: Number of TEAEs by Relationship
Description: The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. Here, number of TEAEs by relationship (related or unrelated to the study drug) are reported.
Time Frame: Day 1 through end of study (Day 24)
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Number; unit: Events
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Events
  Related | 125 | 94
  Unrelated | 9 | 8

22. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Vital Signs
Description: Number of participants with clinically significant abnormal vital signs are reported. Abnormal clinical vital signs are defined as any abnormal finding in the vital sign parameters (blood pressure, heart rate, and oral temperature).
Time Frame: Screening (Day -30 to -3) through Day 24 (end of study)
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Participants | 0 | 0

23. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiograms (ECGs)
Description: Number of participants with clinically significant abnormal ECGs are reported. Abnormal clinical ECG parameters are defined as any abnormal finding during analysis of 12-lead safety ECGs, 12-lead digital ECGs, and ECG telemetry.
Time Frame: Screening (Day -30 to -3) through end of study (Day 24)
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Participants | 2 | 1

24. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Values
Description: Number of participants with clinically significant abnormal laboratory values are reported. Abnormal clinical laboratory parameters are defined as any abnormal finding during analysis of hematology, clinical chemistry, coagulation, and urinalysis.
Time Frame: Screening (Day -30 to Day -3) through end of study (Day 24)
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Participants | 0 | 0

25. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Physical Examination Findings
Description: Number of participants with clinically significant abnormal physical examination findings are reported. The physical examination included a general review of the following body systems (at minimum): head and neck, cardiovascular, respiratory, gastrointestinal, brief neurological and general appearance, unless a symptom oriented physical exam is indicated.
Time Frame: Screening (Day -30 to Day -3) through end of study (Day 24)
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Participants | 0 | 0

26. Secondary Outcome: Number of Participants With Clinically Significant Neurological Examinations Findings
Description: Number of participants with clinically significant neurological examinations findings are reported. Neurological examinations included assessments of basic mental status, cranial nerves, motor function, reflexes, sensation, proprioception, coordination, and gait.
Time Frame: Screening (Day -30 to Day -3) through end of study (Day 24)
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Participants | 0 | 0

27. Secondary Outcome: Number of Participants With Suicidal Ideation or Behaviors Per Columbia-Suicide Severity Rating Scale (C-SSRS) Assessments
Description: The C-SSRS is a suicidal ideation and behavior rating scale with yes/no responses. Items 1-5 rates an individual's degree of suicidal ideation on a 0 (wish to be dead) to 5 (active suicidal ideation with specific plan and intent and behaviors) scale. C-SSRS outcomes are categories and have binary responses (yes/no). Suicidal ideation is considered when the participant responds a 'yes' to any one of the five suicidal ideation questions (Categories 1-5) on the C-SSRS at any time during treatment. Items 6-10 of C-SSRS rates suicidal behavior where outcome is a simple yes/no response. Suicidal behavior was considered if participant answers a 'yes' to any one of the five suicidal behavior questions (Categories 6-10) on C-SSRS at any time during treatment. Number of participants with suicidal behavior and ideation per C-SSRS assessments are reported.
Time Frame: Screening (Day -30 to Day -3) through end of study (Day 24)
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Participants
  Suicidal Ideation | 0 | 0
  Suicidal Behaviours | 0 | 0

28. Secondary Outcome: Number of Participants With Type of Medical Intervention Used for Each Event of Significantly Increased EtCO2, Reduced SpO2, or RR
Description: Number of participants with type of medical intervention used for each event of significantly increased EtCO2, reduced SpO2, or RR are reported.
Time Frame: Screening (Day -30 to Day -3) through end of study (Day 24)
Population: The safety population included all participants who received at least 1 dose of morphine.
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Participants | 0 | 0

29. Secondary Outcome: Maximum Observed Concentration (Cmax) of Morphine and Its Metabolites
Description: The Cmax of morphine and its metabolites (morphine-3-glucuronide and morphine-6-glucuronide) are reported.
Time Frame: Day 1: predose, 0.08, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 36 hours postdose and Day 15: predose, 0.08, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 hours postdose, and additionally 48 hours postdose for morphine metabolites
Population: Pharmacokinetic (PK) population included all participants in the safety population who received at least 1 dose of morphine or AZD4041 and have at least 1 PK concentration after dosing. Number analyzed (n) denotes those participants who had adequate plasma samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
ng/mL
  Morphine (Day 1) | 96.24 (22.07) | 95.51 (16.95)
  Morphine (Day 15): number analyzed (Participants) | 25 | 13
  Morphine (Day 15) | 88.32 (24.14) | 88.54 (20.74)
  Morphine-3-glucuronide (Day 1) | 313.7 (25.54) | 352.9 (14.03)
  Morphine-3-glucuronide (Day 15): number analyzed (Participants) | 25 | 13
  Morphine-3-glucuronide (Day 15) | 291.0 (23.34) | 300.8 (10.58)
  Morphine-6-glucuronide (Day 1) | 56.40 (21.46) | 64.44 (10.60)
  Morphine-6-glucuronide (Day 15): number analyzed (Participants) | 25 | 13
  Morphine-6-glucuronide (Day 15) | 53.54 (19.06) | 59.88 (12.96)

30. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of Morphine and Its Metabolites
Description: The Tmax of morphine and its metabolites (morphine-3-glucuronide and morphine-6-glucuronide) are reported.
Time Frame: as for outcome 29
Population: PK population included all participants in the safety population who received at least 1 dose of morphine or AZD4041 and have at least 1 PK concentration after dosing. Number analyzed (n) denotes those participants who had adequate plasma samples.
Measure: Median (Full Range); unit: Hour
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Hour
  Morphine (Day 1) | 0.08 [0.08 to 0.10] | 0.08 [0.08 to 0.08]
  Morphine (Day 15): number analyzed (Participants) | 25 | 13
  Morphine (Day 15) | 0.08 [0.08 to 0.10] | 0.08 [0.08 to 0.17]
  Morphine-3-glucuronide (Day 1) | 0.25 [0.08 to 1.00] | 0.25 [0.08 to 0.53]
  Morphine-3-glucuronide (Day 15): number analyzed (Participants) | 25 | 13
  Morphine-3-glucuronide (Day 15) | 0.27 [0.08 to 1.03] | 0.27 [0.08 to 1.02]
  Morphine-6-glucuronide (Day 1) | 0.76 [0.25 to 1.50] | 0.50 [0.25 to 1.00]
  Morphine-6-glucuronide (Day 15): number analyzed (Participants) | 25 | 13
  Morphine-6-glucuronide (Day 15) | 1.00 [0.25 to 1.50] | 0.50 [0.28 to 1.50]

31. Secondary Outcome: Area Under Plasma Concentration-time Curve From Zero to the Last Quantifiable Concentration (AUC0-t) of Morphine and Its Metabolites
Description: The AUC0-t of morphine and its metabolites (morphine-3-glucuronide and morphine-6-glucuronide) are reported.
Time Frame: as for outcome 29
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
h*ng/mL
  Morphine (Day 1) | 132.5 (26.78) | 124.5 (23.59)
  Morphine (Day 15): number analyzed (Participants) | 25 | 13
  Morphine (Day 15) | 135.5 (29.08) | 128.2 (17.33)
  Morphine-3-glucuronide (Day 1) | 1996 (18.55) | 2067 (15.21)
  Morphine-3-glucuronide (Day 15): number analyzed (Participants) | 25 | 13
  Morphine-3-glucuronide (Day 15) | 2120 (19.43) | 2194 (15.11)
  Morphine-6-glucuronide (Day 1) | 315.3 (17.76) | 342.0 (18.68)
  Morphine-6-glucuronide (Day 15): number analyzed (Participants) | 25 | 13
  Morphine-6-glucuronide (Day 15) | 342.7 (16.45) | 380.3 (18.66)

32. Secondary Outcome: Area Under Plasma Concentration-time Curve Extrapolated to Infinity (AUC0-∞) of Morphine and Its Metabolites
Description: The (AUC0-∞) of morphine and its metabolites (morphine-3-glucuronide and morphine-6-glucuronide) are reported.
Time Frame: as for outcome 29
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
h*ng/mL
  Morphine (Day 1) | 140.5 (26.30) | 133.8 (21.19)
  Morphine (Day 15): number analyzed (Participants) | 25 | 13
  Morphine (Day 15) | 142.6 (28.33) | 140.8 (17.87)
  Morphine-3-glucuronide (Day 1) | 2259 (20.29) | 2404 (17.43)
  Morphine-3-glucuronide (Day 15): number analyzed (Participants) | 25 | 13
  Morphine-3-glucuronide (Day 15) | 2284 (17.84) | 2363 (15.32)
  Morphine-6-glucuronide (Day 1) | 372.6 (48.69) | 389.4 (17.13)
  Morphine-6-glucuronide (Day 15): number analyzed (Participants) | 25 | 13
  Morphine-6-glucuronide (Day 15) | 371.2 (16.37) | 408.3 (19.38)

33. Secondary Outcome: Terminal Elimination Half-life (t1/2λz) of Morphine and Its Metabolites
Description: The t1/2λz of morphine and its metabolites (morphine-3-glucuronide and morphine-6-glucuronide) are reported.
Time Frame: as for outcome 29
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Hour
  Morphine (Day 1) | 3.131 (49.58) | 3.493 (53.29)
  Morphine (Day 15): number analyzed (Participants) | 25 | 13
  Morphine (Day 15) | 3.090 (32.23) | 4.483 (109.0)
  Morphine-3-glucuronide (Day 1) | 10.04 (62.79) | 11.37 (46.87)
  Morphine-3-glucuronide (Day 15): number analyzed (Participants) | 25 | 13
  Morphine-3-glucuronide (Day 15) | 11.13 (40.00) | 12.39 (24.99)
  Morphine-6-glucuronide (Day 1) | 10.16 (118.2) | 10.38 (51.10)
  Morphine-6-glucuronide (Day 15): number analyzed (Participants) | 25 | 13
  Morphine-6-glucuronide (Day 15) | 10.82 (34.77) | 12.27 (32.34)

34. Secondary Outcome: Time of Last Quantifiable Concentration (Tlast) of Morphine and Its Metabolites
Description: The tlast of morphine and its metabolites (morphine-3-glucuronide and morphine-6-glucuronide) are reported.
Time Frame: as for outcome 29
Population: as for outcome 30
Measure: Median (Full Range); unit: Hours
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Hours
  Morphine (Day 1) | 12.00 [8.00 to 36.00] | 12.00 [8.00 to 24.00]
  Morphine (Day 15): number analyzed (Participants) | 25 | 13
  Morphine (Day 15) | 12.00 [8.00 to 24.10] | 12.00 [8.00 to 24.00]
  Morphine-3-glucuronide (Day 1) | 36.00 [12.00 to 36.10] | 36.00 [24.00 to 36.15]
  Morphine-3-glucuronide (Day 15): number analyzed (Participants) | 25 | 13
  Morphine-3-glucuronide (Day 15) | 48.00 [24.00 to 48.10] | 36.00 [36.00 to 48.00]
  Morphine-6-glucuronide (Day 1) | 36.00 [12.00 to 36.10] | 36.00 [24.00 to 36.15]
  Morphine-6-glucuronide (Day 15): number analyzed (Participants) | 25 | 13
  Morphine-6-glucuronide (Day 15) | 36.03 [24.00 to 48.10] | 36.00 [36.00 to 48.00]

35. Secondary Outcome: Total Body Clearance (CL) of Morphine
Description: The CL of morphine are reported.
Time Frame: as for outcome 29
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
L/h
  Day 1 | 142.4 (26.30) | 149.4 (21.19)
  Day 15: number analyzed (Participants) | 25 | 13
  Day 15 | 140.2 (28.33) | 142.0 (17.87)

36. Secondary Outcome: Volume of Distribution Based on the Terminal Phase (Vz) of Morphine
Description: The Vz of morphine are reported.
Time Frame: as for outcome 29
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
Liter
  Day 1 | 643.2 (41.23) | 753.0 (55.77)
  Day 15: number analyzed (Participants) | 25 | 13
  Day 15 | 625.1 (36.38) | 918.5 (97.58)

37. Secondary Outcome: Maximum Observed Concentration at Steady-state (Cmax,ss) of AZD4041
Description: The Cmax,ss of AZD4041 are reported.
Time Frame: Day 8: predose, 0.08, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose and Day 15: predose, 0.08, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose
Population: PK population included all participants in the safety population who received at least 1 dose of morphine or AZD4041 and have at least 1 PK concentration after dosing. Number of participants analyzed (N) denotes those participants who received at least one dose of AZD4041.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041
Number analyzed (Participants) | 25
ng/mL
  Day 8 | 717.8 (23.95)
  Day 15 | 660.7 (22.14)

38. Secondary Outcome: Time to Reach Maximum Observed Concentration at Steady State (Tmax,ss) of AZD4041
Description: The tmax,ss of AZD4041 are reported.
Time Frame: as for outcome 37
Population: as for outcome 37
Measure: Median (Full Range); unit: Hour
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041
Number analyzed (Participants) | 25
Hour
  Day 8 | 0.50 [0.25 to 1.50]
  Day 15 | 1.57 [0.23 to 7.98]

39. Secondary Outcome: Area Under Plasma Concentration-time Curve Over a Dosing Interval (AUCτ) of AZD4041
Description: The AUCτ of AZD4041 are reported.
Time Frame: as for outcome 37
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041
Number analyzed (Participants) | 25
h*ng/mL
  Day 8 | 7114 (31.15)
  Day 15 | 7711 (28.34)

40. Secondary Outcome: Terminal Elimination Half-life (t1/2λz) of AZD4041
Description: The t1/2λz of AZD4041 are reported.
Time Frame: as for outcome 37
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041
Number analyzed (Participants) | 25
Hour
  Day 8 | 14.44 (63.21)
  Day 15 | 12.14 (39.71)

41. Secondary Outcome: Average Concentration Over a Dosing Interval (Cav) of AZD4041
Description: The Cav of AZD4041 are reported.
Time Frame: as for outcome 37
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041
Number analyzed (Participants) | 25
ng/mL
  Day 8 | 296.4 (31.15)
  Day 15 | 321.3 (28.34)

42. Secondary Outcome: Apparent Total Body Clearance at Steady State (CLss/F) of AZD4041
Description: The CLss/F of AZD4041 are reported.
Time Frame: as for outcome 37
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041
Number analyzed (Participants) | 25
L/h
  Day 8 | 3.514 (31.15)
  Day 15 | 3.242 (28.34)

43. Secondary Outcome: Apparent Volume of Distribution at Steady State Based on the Terminal Phase (Vzss/F) of AZD4041
Description: The Vzss/F of AZD4041 are reported
Time Frame: as for outcome 37
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041
Number analyzed (Participants) | 25
Liter
  Day 8 | 73.19 (57.65)
  Day 15 | 56.79 (37.29)

44. Secondary Outcome: Observed Lowest Concentration Before the Next Dose is Administered at Steady State (Ctrough,ss) of AZD4041
Description: The Ctrough,ss of AZD4041 are reported.
Time Frame: as for outcome 37
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041
Number analyzed (Participants) | 25
ng/mL
  Day 8 | 133.8 (66.35)
  Day 15 | 149.5 (67.10)

45. Secondary Outcome: Amount of AZD4041 Excreted Unchanged in Urine (Aeτ)
Description: The Aeτ of AZD4041 is reported.
Time Frame: Day 15: Predose spot collection, 0 to 6 hours, 6 to 12 hours, 12 to 24 hours, 24 to 48 hours, and 48 to 72 hours postdose
Population: PK population included all participants in the safety population who received at least 1 dose of morphine or AZD4041 and have at least 1 PK concentration after dosing. Number of participants analyzed (N) denotes those participants who received at least one dose of AZD4041 and who were evaluable at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041
Number analyzed (Participants) | 15
ng | 390400 (63.03)

46. Secondary Outcome: Apparent Fraction of AZD4041 Excreted Unchanged in Urine (Feτ/F)
Description: The Feτ/F of AZD4041 is reported.
Time Frame: as for outcome 45
Population: as for outcome 45
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041
Number analyzed (Participants) | 15
Percentage | 1.562 (63.03)

47. Secondary Outcome: Renal Clearance (CLR) of AZD4041
Description: The CLR of AZD4041 is reported.
Time Frame: as for outcome 45
Population: as for outcome 45
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041
Number analyzed (Participants) | 15
L/h | 0.04757 (78.33)

48. Secondary Outcome: Terminal Elimination Half-life (t1/2) of AZD4041
Description: The t1/2 of AZD4041 is reported.
Time Frame: as for outcome 45
Population: as for outcome 37
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041
Number analyzed (Participants) | 22
Hour | 14.48 (111.7)

49. Secondary Outcome: Plasma Concentration of Morphine Over Time
Description: Plasma concentration of morphine over time was reported.
Time Frame: Day 1: predose, 0.08, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, and 36 hours postdose and Day 15: predose, 0.08, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 hours postdose
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
ng/mL
  Day 1 (Predose) | NA (NA) — Data was not reported as the value was below the lower limit of quantification. | NA (NA) — Data was not reported as the value was below the lower limit of quantification.
  Day 1 (0.08 hour) | 96.24 (22.1) | 95.51 (16.9)
  Day 1 (0.25 hour) | 57.04 (23.9) | 54.16 (20.8)
  Day 1 (0.5 hour) | 40.89 (25.5) | 38.50 (22.8)
  Day 1 (1 hour) | 29.42 (29.8) | 26.58 (22.9)
  Day 1 (1.5 hour) | 25.13 (25.3) | 21.07 (24.7)
  Day 1 (2 hour) | 19.43 (25.0) | 17.24 (27.6)
  Day 1 (3 hour) | 14.00 (24.2) | 11.82 (33.9)
  Day 1 (4 hour) | 9.92 (27.7) | 9.50 (30.0)
  Day 1 (6 hour) | 4.99 (33.6) | 4.77 (35.4)
  Day 1 (8 hour) | 3.05 (31.1) | 2.99 (33.7)
  Day 1 (12 hour): number analyzed (Participants) | 24 | 15
  Day 1 (12 hour) | 1.21 (19.1) | 1.32 (25.6)
  Day 1 (24 hour): number analyzed (Participants) | 24 | 14
  Day 1 (24 hour) | NA (NA) — Data was not reported as the value was below the lower limit of quantification. | NA (NA) — Data was not reported as the value was below the lower limit of quantification.
  Day 1 (36 hour): number analyzed (Participants) | 25 | 13
  Day 1 (36 hour) | NA (NA) — Data was not reported as the value was below the lower limit of quantification. | NA (NA) — Data was not reported as the value was below the lower limit of quantification.
  Day 15 (predose): number analyzed (Participants) | 25 | 12
  Day 15 (predose) | NA (NA) — Data was not reported as the value was below the lower limit of quantification. | NA (NA) — Data was not reported as the value was below the lower limit of quantification.
  Day 15 (0.08 hour): number analyzed (Participants) | 25 | 13
  Day 15 (0.08 hour) | 88.32 (24.1) | 88.54 (20.7)
  Day 15 (0.25 hour): number analyzed (Participants) | 25 | 13
  Day 15 (0.25 hour) | 56.83 (24.9) | 53.14 (22.4)
  Day 15 (0.5 hour): number analyzed (Participants) | 25 | 13
  Day 15 (0.5 hour) | 39.88 (29.3) | 38.55 (25.0)
  Day 15 (1 hour): number analyzed (Participants) | 25 | 13
  Day 15 (1 hour) | 30.09 (33.0) | 27.00 (22.1)
  Day 15 (1.5 hour): number analyzed (Participants) | 25 | 13
  Day 15 (1.5 hour) | 24.31 (28.5) | 22.00 (18.0)
  Day 15 (2 hour): number analyzed (Participants) | 25 | 13
  Day 15 (2 hour) | 20.54 (31.2) | 18.09 (21.6)
  Day 15 (3 hour): number analyzed (Participants) | 25 | 13
  Day 15 (3 hour) | 14.16 (29.1) | 13.99 (19.6)
  Day 15 (4 hour): number analyzed (Participants) | 25 | 13
  Day 15 (4 hour) | 10.74 (33.5) | 10.00 (23.6)
  Day 15 (6 hour): number analyzed (Participants) | 25 | 13
  Day 15 (6 hour) | 5.06 (41.5) | 4.87 (35.8)
  Day 15 (8 hour): number analyzed (Participants) | 25 | 13
  Day 15 (8 hour) | 2.85 (34.4) | 2.93 (34.0)
  Day 15 (12 hour): number analyzed (Participants) | 24 | 12
  Day 15 (12 hour) | 1.42 (30.0) | 1.36 (26.1)
  Day 15 (24 hour): number analyzed (Participants) | 24 | 12
  Day 15 (24 hour) | NA (NA) — Data was not reported as the value was below the lower limit of quantification. | NA (NA) — Data was not reported as the value was below the lower limit of quantification.
  Day 15 (36 hour): number analyzed (Participants) | 25 | 13
  Day 15 (36 hour) | NA (NA) — Data was not reported as the value was below the lower limit of quantification. | NA (NA) — Data was not reported as the value was below the lower limit of quantification.

50. Secondary Outcome: Plasma Concentration of Morphine-3-glucuronide Over Time
Description: Plasma concentration of morphine-3-glucuronide over time are reported.
Time Frame: as for outcome 29
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
ng/mL
  Day 1 (predose) | NA (NA) — Data was not reported as the value was below the lower limit of quantification. | NA (NA) — Data was not reported as the value was below the lower limit of quantification.
  Day 1 (0.08 hours) | 261.17 (42.9) | 330.85 (16.9)
  Day 1 (0.25 hours) | 287.69 (28.3) | 336.02 (12.7)
  Day 1 (0.5 hours) | 282.31 (27.1) | 311.44 (10.9)
  Day 1 (1 hours) | 257.89 (27.7) | 276.48 (14.7)
  Day 1 (1.5 hours) | 244.91 (22.4) | 247.20 (15.5)
  Day 1 (2 hours) | 222.77 (20.1) | 215.93 (18.5)
  Day 1 (3 hours) | 179.81 (24.0) | 163.04 (39.6)
  Day 1 (4 hours) | 146.71 (24.6) | 146.83 (19.0)
  Day 1 (6 hours) | 97.80 (24.3) | 92.21 (21.7)
  Day 1 (8 hours) | 65.29 (23.1) | 57.07 (30.3)
  Day 1 (12 hours) | 30.21 (44.6) | 35.03 (43.0)
  Day 1 (24 hours): number analyzed (Participants) | 25 | 15
  Day 1 (24 hours) | 23.17 (32.8) | 27.71 (32.8)
  Day 1 (36 hours): number analyzed (Participants) | 25 | 13
  Day 1 (36 hours) | 12.53 (48.8) | 14.19 (39.6)
  Day 15 (predose): number analyzed (Participants) | 25 | 12
  Day 15 (predose) | NA (NA) — Data was not reported as the value was below the lower limit of quantification. | NA (NA) — Data was not reported as the value was below the lower limit of quantification.
  Day 15 (0.08 hours): number analyzed (Participants) | 25 | 13
  Day 15 (0.08 hours) | 235.04 (42.8) | 255.36 (31.2)
  Day 15 (0.25 hours): number analyzed (Participants) | 25 | 13
  Day 15 (0.25 hours) | 262.41 (34.6) | 289.85 (14.2)
  Day 15 (0.5 hours): number analyzed (Participants) | 25 | 13
  Day 15 (0.5 hours) | 263.96 (34.7) | 278.58 (16.7)
  Day 15 (1 hours): number analyzed (Participants) | 25 | 13
  Day 15 (1 hours) | 254.13 (21.3) | 264.39 (11.8)
  Day 15 (1.5 hours): number analyzed (Participants) | 25 | 13
  Day 15 (1.5 hours) | 234.80 (19.5) | 243.99 (13.7)
  Day 15 (2 hours): number analyzed (Participants) | 25 | 13
  Day 15 (2 hours) | 213.71 (19.6) | 218.39 (14.8)
  Day 15 (3 hours): number analyzed (Participants) | 25 | 13
  Day 15 (3 hours) | 176.05 (22.2) | 179.70 (16.0)
  Day 15 (4 hours): number analyzed (Participants) | 25 | 13
  Day 15 (4 hours) | 144.41 (24.8) | 145.37 (19.5)
  Day 15 (6 hours): number analyzed (Participants) | 25 | 13
  Day 15 (6 hours) | 91.78 (41.4) | 91.87 (15.8)
  Day 15 (8 hours): number analyzed (Participants) | 25 | 13
  Day 15 (8 hours) | 62.28 (28.5) | 59.38 (21.4)
  Day 15 (12 hours): number analyzed (Participants) | 25 | 13
  Day 15 (12 hours) | 39.26 (34.7) | 30.01 (47.6)
  Day 15 (24 hours): number analyzed (Participants) | 25 | 13
  Day 15 (24 hours) | 24.87 (31.9) | 27.49 (24.3)
  Day 15 (36 hours): number analyzed (Participants) | 25 | 13
  Day 15 (36 hours) | 11.78 (53.7) | 16.90 (26.2)
  Day 15 (48 hours): number analyzed (Participants) | 25 | 13
  Day 15 (48 hours) | 6.76 (38.0) | 8.40 (30.5)

51. Secondary Outcome: Plasma Concentration of Morphine-6-glucuronide Over Time
Description: Plasma concentration of morphine-6-glucuronide over time are reported.
Time Frame: as for outcome 29
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
Number analyzed (Participants) | 26 | 15
ng/mL
  Day 1 (predose) | NA (NA) — Data was not reported as the value was below the lower limit of quantification. | NA (NA) — Data was not reported as the value was below the lower limit of quantification.
  Day 1 (0.08 hours) | 22.52 (53.0) | 32.79 (23.4)
  Day 1 (0.25 hours) | 42.25 (35.8) | 56.30 (17.1)
  Day 1 (0.5 hours) | 51.95 (27.4) | 62.02 (8.9)
  Day 1 (1 hours) | 51.22 (24.5) | 57.49 (16.2)
  Day 1 (1.5 hours) | 46.95 (17.7) | 50.15 (13.6)
  Day 1 (2 hours) | 41.86 (16.0) | 42.36 (22.5)
  Day 1 (3 hours) | 31.64 (18.3) | 29.23 (37.9)
  Day 1 (4 hours) | 23.97 (20.3) | 25.24 (20.2)
  Day 1 (6 hours) | 14.95 (23.5) | 14.55 (24.0)
  Day 1 (8 hours) | 9.05 (22.3) | 8.32 (32.7)
  Day 1 (12 hours) | 3.83 (41.4) | 4.88 (46.8)
  Day 1 (24 hours): number analyzed (Participants) | 25 | 15
  Day 1 (24 hours) | 3.45 (43.1) | 4.30 (37.1)
  Day 1 (36 hours): number analyzed (Participants) | 25 | 13
  Day 1 (36 hours) | 1.76 (45.5) | 1.91 (40.9)
  Day 15 (predose): number analyzed (Participants) | 25 | 12
  Day 15 (predose) | NA (NA) — Data was not reported as the value was below the lower limit of quantification. | NA (NA) — Data was not reported as the value was below the lower limit of quantification.
  Day 15 (0.08 hours): number analyzed (Participants) | 25 | 13
  Day 15 (0.08 hours) | 20.40 (55.9) | 23.45 (44.8)
  Day 15 (0.25 hours): number analyzed (Participants) | 25 | 13
  Day 15 (0.25 hours) | 37.25 (43.5) | 46.21 (21.8)
  Day 15 (0.5 hours): number analyzed (Participants) | 25 | 13
  Day 15 (0.5 hours) | 48.42 (34.5) | 56.18 (19.4)
  Day 15 (1 hours): number analyzed (Participants) | 25 | 13
  Day 15 (1 hours) | 51.86 (18.6) | 57.32 (13.0)
  Day 15 (1.5 hours): number analyzed (Participants) | 25 | 13
  Day 15 (1.5 hours) | 47.25 (15.7) | 52.46 (14.1)
  Day 15 (2 hours): number analyzed (Participants) | 25 | 13
  Day 15 (2 hours) | 41.51 (16.4) | 46.16 (15.5)
  Day 15 (3 hours): number analyzed (Participants) | 25 | 13
  Day 15 (3 hours) | 32.10 (14.8) | 34.90 (17.5)
  Day 15 (4 hours): number analyzed (Participants) | 25 | 13
  Day 15 (4 hours) | 25.57 (15.6) | 26.76 (19.0)
  Day 15 (6 hours): number analyzed (Participants) | 25 | 13
  Day 15 (6 hours) | 14.39 (34.7) | 15.20 (20.3)
  Day 15 (8 hours): number analyzed (Participants) | 25 | 13
  Day 15 (8 hours) | 8.93 (23.6) | 9.15 (25.8)
  Day 15 (12 hours): number analyzed (Participants) | 25 | 13
  Day 15 (12 hours) | 5.57 (37.0) | 4.39 (54.5)
  Day 15 (24 hours): number analyzed (Participants) | 25 | 13
  Day 15 (24 hours) | 3.84 (34.4) | 4.43 (32.2)
  Day 15 (36 hours): number analyzed (Participants) | 25 | 13
  Day 15 (36 hours) | 1.73 (47.3) | 2.51 (27.0)
  Day 15 (48 hours): number analyzed (Participants) | 25 | 13
  Day 15 (48 hours) | NA (NA) — Data was not reported as the value was below the lower limit of quantification. | 1.34 (33.5)

52. Secondary Outcome: Plasma Concentration of AZD4041 Over Time
Description: Plasma concentration of AZD4041 over time are reported.
Time Frame: Day 8: predose, 0.08, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose, and Day 15: predose, 0.08, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours postdose
Population: PK population included all participants in the safety population who received at least 1 dose of morphine or AZD4041 and have at least 1 PK concentration after dosing. Number of participants analyzed (N) denotes those participants who received at least one dose of AZD4041. Number analyzed (n) denotes those participants who had adequate plasma samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041
Number analyzed (Participants) | 25
ng/mL
  Day 8 (predose) | 133.83 (66.4)
  Day 8 (0.08 hours) | 186.27 (47.3)
  Day 8 (0.25 hours) | 435.07 (44.6)
  Day 8 (0.5 hours) | 690.91 (28.7)
  Day 8 (1 hours) | 623.75 (28.5)
  Day 8 (1.5 hours) | 602.16 (32.6)
  Day 8 (2 hours) | 576.78 (25.2)
  Day 8 (3 hours) | 531.67 (29.9)
  Day 8 (4 hours) | 508.05 (30.2)
  Day 8 (6 hours) | 353.26 (33.5)
  Day 8 (8 hours) | 327.88 (34.6)
  Day 8 (12 hours) | 227.32 (41.2)
  Day 8 (24 hours) | 136.56 (57.7)
  Day 15 (predose) | 149.54 (67.1)
  Day 15 (0.08 hours) | 192.53 (53.2)
  Day 15 (0.25 hours) | 369.16 (52.5)
  Day 15 (0.5 hours) | 467.16 (45.1)
  Day 15 (1 hours) | 504.23 (33.6)
  Day 15 (1.5 hours) | 546.10 (35.0)
  Day 15 (2 hours) | 523.23 (33.4)
  Day 15 (3 hours) | 566.76 (23.2)
  Day 15 (4 hours) | 524.01 (34.6)
  Day 15 (6 hours) | 432.55 (29.7)
  Day 15 (8 hours) | 380.48 (33.5)
  Day 15 (12 hours): number analyzed (Participants) | 24
  Day 15 (12 hours) | 264.56 (39.4)
  Day 15 (24 hours) | 157.21 (53.4)
  Day 15 (36 hours) | 54.33 (94.5)
  Day 15 (48 hours) | 33.77 (133.2)
  Day 15 (72 hours) | 7.97 (240.0)

ADVERSE EVENTS:
Time Frame: Day 1 through end of study (Day 24)
Description: The safety population included all participants who received at least 1 dose of morphine.
Arm/Group | Morphine Then AZD4041 Then Morphine + AZD4041 | Morphine Then Placebo Then Morphine + Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/15
Other Adverse Events (participants affected / at risk) | 26/26 | 14/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine Then AZD4041 Then Morphine + AZD4041 (N=26) | Morphine Then Placebo Then Morphine + Placebo (N=15)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (9) | 6 (11)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (11) | 6 (11)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 4 (5) | 2 (3)
Feeling abnormal (General disorders) | 4 (4) | 3 (4)
Feeling hot (General disorders) | 12 (14) | 7 (10)
Feeling of relaxation (General disorders) | 3 (3) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
End-tidal Co2 increased (Investigations) | 2 (2) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (6) | 1 (1)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (5) | 5 (6)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 3 (3) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 12 (14) | 7 (8)
Euphoric mood (Psychiatric disorders) | 12 (17) | 12 (18)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (11) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 2 (2)
Lacrimation increased (Eye disorders) | 1 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT05587998/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT05587998/SAP_001.pdf